CLINICAL TRIAL: NCT05267327
Title: A Prospective Post-Marketing Observational Safety Study of Verzenios® (Abemaciclib) Among Breast Cancer Patients in China
Brief Title: A Prospective Post-Marketing Observational Safety Study of Verzenios® (Abemaciclib) Among Breast Cancer Patients in China Verzenios® (Abemaciclib) Among Breast
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: I3Y-MC-B009
Record Dates: First submitted 2022-02-28; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: The Incidence of AEs and SAEs Receiving Verzenios® Over a Period of Approximately 24 Weeks

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 104 Weeks
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Verzenios — Study drug is Verzenios, it is an observational study.

SUMMARY:
This PMSS is a single-country, prospective, observational study primarily designed to estimate the incidence of AEs and SAEs among Chinese patients with breast cancer after receiving Verzenios® over a period of approximately 24 weeks in a routine clinical practice. According to the pivotal studies (MONARCH 2, 3 and MONARCH plus), the most frequent treatment-emergent adverse events (TEAEs) generally reported occurred at an early time (within 28 days after treatment initiation) point during treatment (Dickler et al. 2017); hence, each patient enrolled in the study will have the first follow-up visit at 4 ± 1 weeks after the first abemaciclib treatment for regular safety monitoring. Since most reported TEAEs occur within 6 months, patients will return to the clinic after receiving Verzenios for 6 months to carry out the routine effectiveness evaluation in the normal clinical practice setting. The observational duration for primary objective is set as 24 ± 4 weeks. Moreover, the effectiveness related variables including ORR, DCR, EFS rate, and OS rate, if available, will be investigated as the secondary objectives of the study and patients will be followed for 24 ± 4 weeks and up to 2 years (only for EFS rate and OS rate) after initiation of Verzenios. Approximately 30 hospitals across China are planned for participation in this study. This study plans to enroll approximately 1500 patients (detailed in Section 9.5) and both safety and effectiveness of Verzenios will be evaluated. The observation period for each patient will be either until the last Verzenios treatment (if patients discontinue Verzenios before the follow-up duration of 24 weeks for safety and effectiveness [EFS rate and OS rate will be assessed at 52 weeks and 104 weeks], 30 days follow-up will be carried out for safety events), or follow-up discontinuation (for example, death), whichever comes first. Visits will be performed at baseline (baseline visit), 4 weeks (Visit 1), 12 weeks (Visit 2), and 24 weeks (Visit 3) of treatment for safety and effectiveness assessments. Follow-up visits will be performed at 52 weeks (Visit 4) and 104 weeks (Visit 5) of treatment for OS rate assessment.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old at enrolment
* diagnosed with HR-positive, HER2-negative breast cancer
* prescribed with Verzenios by the investigators and started (or planned to start shortly) Verzenios treatment in the routine care of the patient
* provide written consent to the release of their data after being informed of the study.

Exclusion Criteria:

* have been administered Verzenios before study enrollment
* are simultaneously participating in a different study that includes a treatment intervention and/or an investigational drug
* are pregnant or breastfeeding or intend to become pregnant within the duration of the study
* contraindicated for the use of Verzenios according to the China approved label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients (≥18 years old at enrollment) who have been diagnosed with breast cancer, have been prescribed Verzenios in a routine clinical care setting by the investigator, and have provided written consent to release their data after being informed of the study.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The Incidence of AEs and SAEs | 24 Weeks
  The observation period for each patient for AE/SAE

IPD SHARING:
Plan to Share IPD: Undecided